CLINICAL TRIAL: NCT03652870
Title: A Randomised Placebo-Controlled Trial of Escitalopram and Nortriptyline With Standard Psychological Care for Depression in Parkinson's Disease
Brief Title: Antidepressants Trial in Parkinson's Disease
Acronym: ADepT-PD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University College, London (Other)
Collaborators: London North West Healthcare NHS Trust (Other); King's College London (Other); University Hospital Plymouth NHS Trust (Other); NHS Lothian (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 18/0279
Record Dates: First submitted 2018-08-08; First posted 2018-08-29 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Depression; Parkinson Disease
Keywords: Parkinson's Disease
MeSH Terms: conditions — Depression; Parkinson Disease | interventions — Nortriptyline; Escitalopram

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Nortriptyline (Active Comparator): 25mg tablet to be escalated from one tablet per day to a maximum of 4 tablets per day
  Interventions: Drug: Nortriptyline
- Escitalopram (Active Comparator): 5mg tablet to be escalated from one tablet per day to a maximum of 4 tablets per day
  Interventions: Drug: Escitalopram
- Placebo (Placebo Comparator): The placebo tablet consists of lactose and magnesium stearate. One tablet to be escalated from one tablet per day to a maximum of 4 tablets per day
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Nortriptyline — A medication used to treat conditions such as depression
  Other Names: Nortriptyline 25mg
  Arms: Nortriptyline
Drug: Escitalopram — A medication used to treat conditions such as depression
  Other Names: Escitalopram 5mg
  Arms: Escitalopram
Drug: Placebo — Lactose and magnesium stearate tablet to be used as a placebo.
  Other Names: Placebo oral tablet
  Arms: Placebo

SUMMARY:
This is a randomised trial in a NHS setting, comparing the clinical effectiveness and cost-effectiveness of the selective serotonin reuptake inhibitor, escitalopram, and of the tricyclic antidepressant, nortriptyline, to placebo, undertaken in a real-life setting in addition to standard psychological care for the treatment of patients with depression in Parkinson's disease. Participants will be randomly allocated 1:1:1 to receive escitalopram or nortriptyline or placebo.

DETAILED DESCRIPTION:
Parkinson's disease is a progressive neurological disorder that leads to increasing disability and functional decline. Currently no medications have been shown to halt or delay disease progression and one of the most common complications in patients with this diagnosis is depression . Depressive disorders which affects approximately 40% of patients with Parkinson's disease. They are linked to functional impairment, cognitive decline and faster disease progression and are the main determinant of poor quality of life in Parkinson's disease. Psychological therapies are used via standard access to appropriate psychological services in the NHS, but often antidepressant medications are required. Despite the high incidence of depression in this population, However, no conclusive evidence on appropriate choice of antidepressants in Parkinson's disease exists in the NHS, and the risk of worsening of Parkinsonism and aggravation of non-motor features of Parkinson's disease by antidepressants pose particular challenges in this population.

Based on the previous evidence from small trials, the hypothesis is that both selective serotonin reuptake inhibitors and tricyclic antidepressants are effective compared to placebo and the difference in efficacy between tricyclic antidepressants and selective serotonin reuptake inhibitors is likely to be small, but that the tolerability of selective serotonin reuptake inhibitors is higher in this population than that of tricyclic antidepressants due to the rate of adverse effects. The trial is designed to have statistical power to identify effects that are clinically important and slightly smaller than the pooled effects identified in the existing trials of selective serotonin reuptake inhibitors.

Escitalopram is an selective serotonin reuptake inhibitor similar to citalopram, the most widely used selective serotonin reuptake inhibitor in the UK. Both citalopram and escitalopram, the S-enantiomer, are now off-patent with comparable costs and similar trial results. Until recently, escitalopram has been used less commonly in the NHS as because it was more expensive. However comparative trial data in major depression (including non-industry funded research) suggest that escitalopram is more effective than citalopram with similar or lower rates of side effects, and that it is associated with increased probability of response in trials of older patients with dementia and agitation. In addition, it has been reported that escitalopram has the highest probability of remission and is the most effective and cost-effective pharmacological treatment in a primary care setting.

Amitriptyline is the most widely used tricyclic antidepressants in the UK, but is used predominantly at low doses for pain and insomnia in Parkinson's disease. The side effect profile of amitriptyline makes it poorly tolerated in patients with Parkinson's disease at higher, antidepressant doses. Nortriptyline is a metabolite of amitriptyline. However, unlike amitriptyline it has mainly noradrenergic effects, and weakly blocks dopaminergic reuptake. It also has fewer sedative, α1-blocking and anticholinergic effects than amitriptyline (by a factor of 8). It has been evaluated in multiple trials over several decades and its efficacy and adverse event profile in depressive disorders has been well studied. The trial evidence on tricyclic antidepressants in depression in Parkinson's disease mainly reports on nortriptyline and desipramine (which is not available in the NHS). Whilst nortriptyline has a slightly higher cost than amitriptyline in the NHS, nortriptyline is a more appropriate medication for treatment of depression in this population. In addition, there is accumulating evidence from pre-clinical studies that nortriptyline may delay disease progression in Parkinson's disease.

Patients who meet eligibility criteria at the screening visit will be randomly assigned to receive 52 weeks of double-blind treatment with either escitalopram, or nortriptyline or placebo in a 1-1-1 ratio.

For the first two weeks of double-blind treatment, participants aged 65 years and under will be instructed to take one tablet per day of study drug, containing either 5 mg escitalopram or 25mg nortriptyline or placebo. Thereafter, the daily study medication dosage will be increased by one tablet per day, at two-weekly intervals, to a maximum of four tablets per day unless a subject is experiencing troubling side effects. In those aged over 65 years and in those with hepatic impairment the dose will be increased to two tablets after 2 weeks only, from 5 mg escitalopram to 10mg escitalopram or from 25 nortriptyline to 50mg nortriptyline.

After the primary endpoint at 8 weeks, all participants will continue on the same dose until the study visit at 52 weeks with an intermediate assessment at 26 weeks. Following the study assessment after 52 weeks on medication, the trial drug will be tapered off over 4 weeks in dose reductions of 25 mg for nortriptyline and 5mg for escitalopram every week (4 weeks for participants 65 years or under and 2 weeks for participants aged over 65 years or those with hepatic impairment).

ELIGIBILITY:
Inclusion Criteria:

1. Patients with a diagnosis of idiopathic Parkinson's Disease, based on a history and neurological exam performed by the enrolling investigator with presence of at least two of the three cardinal signs of Parkinson's Disease: rigidity, bradykinesia, and rest tremor with no evidence of diagnostic alternatives. Patients who have been treated with levodopa must have demonstrated a clear response.
2. Aged 18 years old or above
3. Fulfilling diagnostic (DSM-V) criteria for a depressive disorder (i.e., major depressive disorder or persistent depressive disorder) or operationally defined subsyndromal depression (presence of two or more depressive symptoms at threshold or subthreshold levels, at least one of which has to include depressed mood or anhedonia
4. Beck Depression Inventory-II (BDI-II) score ≥14
5. Written informed consent provided
6. Treatment with antiparkinsonian medication is optimised or stable for at least 4 weeks before date of randomisation and there are no plans to change up to primary endpoint (8 weeks).

Exclusion Criteria:

1. Women who are pregnant, breastfeeding or of childbearing potential without effective contraception (hormonal or barrier method of birth control; or abstinence)
2. Patients not able to communicate answers to the self-rating questionnaires
3. Patients with Montreal Cognitive Assessment (MoCA) score <16 or without capacity to consent
4. Treatment with an antidepressant within 4 weeks of enrolment (except for a small dose of amitriptyline up to 50 mg for indications other than depression)
5. Patients with known severe liver failure.
6. Absolute contraindications to escitalopram or nortriptyline. These include:

   1. Patients with known QT-interval prolongation or congenital long QT syndrome.
   2. Recent myocardial infarction (<3 months), any degree of heart block or other cardiac arrhythmias precluding treatment with nortriptyline or escitalopram according to clinical judgement.
7. Medications contraindicated on nortriptyline or escitalopram. These include:

   1. Non-selective and selective irreversible monoamine oxidase inhibitors (MAOIs) within 14 days. However, the antiparkinsonian selective reversible MAO-B inhibitors rasagiline, selegiline and safinamide are not contraindicated.
   2. Concomitant QT prolonging drugs, including domperidone, apomorphine at high doses (single dose or hourly rate of >6mg), certain neuroleptics (not quetiapine or clozapine), quinine, class IA and III antiarrhythmics (amiodarone, dronedarone and disopyramide), the antihistamines astemizole, mizolastine, the antimicrobial agents sparfloxacin, moxifloxacin, erythromycin IV, pentamidine, anti-malarian treatment),and some antiretrovirals.
8. Patients indicating active suicidal ideation or intent on the BDI-II item 9 and who, after clinical review of risk using the standardised Suicide Risk Management Protocol, need to be referred for immediate treatment.
9. Participation in another clinical trial of an investigational medicinal product or device within the last 30 days.
10. Any clinical condition which in the opinion/ clinical judgement of the investigator would make the patient unsuitable for the trial due to safety concerns.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2021-03-05 (Actual); Primary Completion 2023-01-23 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
Depressive symptoms | 8 weeks
  Measured using the Beck Depression Inventory II to assess the severity of depression

SECONDARY OUTCOMES:
Level of depression | 26 and 52 Weeks
  Measured using Beck Depression Inventory II to assess the severity of depression
Severity of depression | 8, 26 and 52 Weeks
  Measured using Patient Health Questionnaire 9 to monitor the severity of depression and response to treatment
Number of patients suffering side effects | 8, 26 and 52 Weeks
  Measured using the Toronto side effects scale which records symptoms specific to depression.
Number of participants suffering side effects | 8, 26 and 52 Weeks
  Measured using reporting of other adverse events not reported on the Toronto side effects scale.
Overall clinical effectiveness | 8, 26 and 52 Weeks
  Measured using the Global Clinical Impression scale - change in health question to rate the severity of the patient's illness.
Anxiety symptoms | 8, 26 and 52 Weeks
  Measured using the Parkinson's Anxiety Scale (PAS) to measure anxiety in patients with Parkinson's disease
Capability | 8, 26 and 52 Weeks
  Measured using ICECAP to measure the patient's capability
Self-rated health score | 8, 26 and 52 Weeks
  Measured using EQ-5D-5L to measure the patients' health score on the day of assessment
Health and social care resource | 8, 26 and 52 Weeks
  Measured using modified Client Service Receipt Inventory (CSRI) to collect information on the whole range of services and supports patients may use
Changes in concomitant medication | 8, 26 and 52 Weeks
  Measured using concomitant medication logs
Motor and non-motor experiences | 8, 26 and 52 Weeks
  Measured using the Movement Disorder Society - Unified Parkinson's Disease Rating Scale to assess both motor and non-motor symptoms associated with Parkinson's disease
Cognitive function | 8, 26 and 52 Weeks
  Measured using Montreal Cognitive Assessment (MoCA) to assess for mild cognitive dysfunction
Levodopa equivalence dose | 8, 26 and 52 Weeks
  Measured using concomitant medication logs to calculate the contribution made by each of the patient's Parkinson's drugs, using, as a common denominator, an estimate of the levodopa equivalent dose
Number of drop outs | 8, 26 and 52 Weeks
  Measured using recruitment logs to determine the number of patients who did not complete the study to the end of study treatment
Carer's self-rated health score | 8, 26 and 52 Weeks
  Measured using EQ-5D-5L to measure the carer' health score on the day of assessment
Carer reported quality of life | 8, 26 and 52 Weeks
  Measured using Carers Quality of Life Questionnaire for Parkinsonism to assess the quality of life of carers of patients with Parkinson's disease

CONTACTS AND LOCATIONS:
Overall Officials: Anette Schrag, Principal Investigator — University College, London
Locations (1):
- Royal Free London NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Schrag A, Carroll C, Lewis G, Serfaty M, Duncan G, Molloy S, Whipps J, McLennan B, Weng JYJ, Hunter RM, Clarke CS, Freemantle N, Embleton-Thirsk A. Effectiveness of Escitalopram and Nortriptyline on Depressive Symptoms in Parkinson's disease: the ADepT-PD RCT pilot. Health Technol Assess. 2025 Nov;29(57):1-78. doi: 10.3310/HFDO7575. PMID 41217862
- [Derived] Schrag A, Carroll C, Duncan G, Molloy S, Grover L, Hunter R, Brown R, Freemantle N, Whipps J, Serfaty MA, Lewis G. Antidepressants Trial in Parkinson's Disease (ADepT-PD): protocol for a randomised placebo-controlled trial on the effectiveness of escitalopram and nortriptyline on depressive symptoms in Parkinson's disease. BMC Neurol. 2022 Dec 12;22(1):474. doi: 10.1186/s12883-022-02988-5. PMID 36510237